CLINICAL TRIAL: NCT00026611
Title: A Multicenter, Double-Blind, Randomized Dose-Response Study of Dryvax Vaccine Against Smallpox in Previously Unvaccinated Adults
Brief Title: A Study of Dryvax Vaccine Against Smallpox in Previously Unvaccinated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: DMID 01-632
Record Dates: First submitted 2001-11-12; First posted 2001-11-13 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-03

CONDITIONS: Smallpox
Keywords: Vaccine prophylaxis
MeSH Terms: conditions — Smallpox | interventions — DryVax vaccine

INTERVENTIONS:
Biological: Dryvax vaccine

SUMMARY:
The purpose of this study is to see how many people respond to a smallpox vaccine when a sore forms where the shot was given.

The world was declared free of smallpox in 1980. General routine vaccinations for smallpox were stopped in the U.S. in 1971. In 1976, the recommendation for routine vaccination of healthcare workers was also discontinued. The only people who presently receive this vaccine are people who work with vaccinia virus or monkeypox virus. Because the world was considered free of smallpox infections, this vaccine was no longer produced; there is a limited supply available in the United States.

Because of the limited amount of Dryvax vaccine (vaccinia virus) against smallpox, this study will look at the ability to dilute the vaccine making more doses available in the event of a smallpox outbreak. The study seeks to characterize a strategy of vaccination against smallpox with various doses of Dryvax, followed by revaccination with the same dose, if required, in volunteers 18-32 years of age with a negative history of smallpox vaccination.

ELIGIBILITY:
Inclusion Criteria:

Patients may be eligible for this study if they:

* Are between 18 and 32 years of age.
* Give written informed consent.
* Are available for follow-up for 2.5 months.
* Have an acceptable medical history by screening evaluation and brief clinical assessment.
* Are HIV-negative.
* Agree to use acceptable contraception and to not get pregnant during the study.

Exclusion Criteria:

Patients may not be eligible for this study if they:

* Have a suppressed immune system.
* Have participated in an HIV vaccine trial.
* Have liver disease, diabetes, or kidney problems.
* Have malignant skin cancer.
* Have autoimmune disease.
* Have used medication that suppresses the immune system.
* Have had psychiatric or medical problems or have job responsibilites that will keep them from participating in the study.
* Use illegal intravenous drugs.
* Have received any live vaccines within 60 days of study start.
* Have used experimental therapies within 30 days before study start.
* Have been vaccinated with certain experimental vaccines.
* Have a vaccination scar but have no record of having a vaccine.
* Have received a smallpox vaccine.
* Have taken blood products or immunoglobulin in the past 6 months.
* Have a fever on the day of vaccination.
* Have certain skin disorders, including eczema, exfoliative skin, lacerations that require stitches or burns larger than 2 x 2 cm.
* Live with, have sexual contact with, or work with anyone who is pregnant, less than a year old, has eczema, has certain skin disorders, has a disease or takes medication that suppresses the immune system.
* Have a condition that, in the opinion of the investigator, might interfere with the study.
* Are allergic to any parts of the vaccine.
* Are allergic to thimerosal, immunoglobulins, cidofovir, or probenecid.
* Are pregnant or breast feeding.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland, Baltimore, Maryland
  - St. Louis University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Frey SE, Couch RB, Tacket CO, Treanor JJ, Wolff M, Newman FK, Atmar RL, Edelman R, Nolan CM, Belshe RB; National Institute of Allergy and Infectious Diseases Smallpox Vaccine Study Group. Clinical responses to undiluted and diluted smallpox vaccine. N Engl J Med. 2002 Apr 25;346(17):1265-74. doi: 10.1056/NEJMoa020534. Epub 2002 Mar 28. PMID 11923490